CLINICAL TRIAL: NCT05277883
Title: The Influence of Lower Extremity and Pelvic Alignment on Accuracy of Hip-Knee-Ankle Radiograph Measurements Before Total Knee Arthroplasty
Brief Title: Influence of Knee Alignment and Pelvis Rotation on Accuracy of Radiograph Measurements Before Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Valdoltra Orthopedic Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Valdoltra - x-ray accuracy
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-12

CONDITIONS: Knee Osteoarthritis
Keywords: knee aligment; total knee arthroplasty; coronal alignment of the lower limb; x-ray accuracy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group: All patients scheduled for a total knee arthroplasty without any previous lower limb deformities or previous hip/knee surgery will be enrolled. A long leg standing x-ray and a CT scan of the lower limb will be obtained for every patient.
  Interventions: Radiation: CT scan

INTERVENTIONS:
Radiation: CT scan — CT of the lower limb

SUMMARY:
The aim of this study is to determine the accuracy of long leg standing X-rays with respect to coronal alignment of the knee.

DETAILED DESCRIPTION:
Long leg standing x-ray is a routine examination to measure the femoral valgus angle before a total knee arthroplasty. Newer studies have shown that coronal leg alignment influences the rotation of the distal femoral part. This rotation might influence the measurements obtained with a long leg standing x-ray.

The primary purpose of this study is to determine whether there is a significant difference between 2D measurements taken on the x-ray and 3D measurements obtained with a CT scan.

ELIGIBILITY:
Inclusion Criteria:

Knee osteoarthritis scheduled for knee arthroplasty

Exclusion Criteria:

* previous leg deformities or surgery that changes alignment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that require primary knee replacement will be enrolled in the study. Patients with prevoius surgery that might had already changed the leg aligment (hip/knee artroplasty, osteotomy) or patients with previous leg deformity are not eligible for the enrolment. Women in reproductive age are also not eligible.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
The angle difference between an x-ray and a CT scan | Before surgery
  The femoral valgus angle, femoral mechanical angle, tibial mechanical angle and hip knee ankle angle are measured separately on the x-ray and on the CT scan. The difference in individual angle is the calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Strahovnik, Principal Investigator — Valdoltra Orthopaedic Hospital
Locations (1):
- Orthopaedic Hospital Valdoltra, Ankaran, Slovenia, Slovenia

IPD SHARING:
Plan to Share IPD: No